CLINICAL TRIAL: NCT01405703
Title: Percutaneous Versus Open Plate Fixation of Diaphyseal Clavicle Fractures
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Kubiak, M.D., University of Utah
Other Study IDs: 36814
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Clavicle Fracture
Keywords: Clavicle Fractures; Numbness; Percutaneous plate fixation; open plate fixation; incision related numbness; union rates; subjective; questionnaire based outcomes; Diaphyseal
MeSH Terms: conditions — Hypesthesia | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- percuataneous plate fixation: an approach with three small longitudinal incisions
  Interventions: Other: xrays
- open plate fixation: large transverse incision
  Interventions: Other: xrays

INTERVENTIONS:
Other: xrays — xrays from 2 week postop to 5 year postop

SUMMARY:
This is a prospective, level II evidence comparison between two cohorts. This study is designed to compare the percutaneous versus open approach for plate fixation of diaphyseal clavicle fractures. This study includes questionnaires and measurements that will collect data on incision-related numbness, union rates, overall outcomes, complication rates of the two methods, infection rates, and overall satisfaction. The surgical procedure, all radiographs and follow-up visits to a minimum of one year are the principle investigators (PI's) standard of care for this injury. Measurements and questionnaires are related to the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* displaced (i.e., no cortical contact of fracture ends on two xray view) diaphyseal clavicle fracture
* fracture pattern amenable to plate fixation
* neurologic injury requiring open reduction
* open clavicle fracture
* clavicle nonunion (defined as an absence of radiographic bony union in the presence of neurologic, cosmetic, or functional complaints at six months duration
* symptomatic malunion (defined as a healed, but shortened or angulated fracture in the presence of neurologic, cosmetic, or functional complaints)
* clavicle fracture associated with a scapular of humeral fracture (floating shoulder)

Exclusion Criteria:

* a nondisplaced or minimally displaced closed, neurovascularly intact clavicle fracture
* fracture of the medial or lateral end of the clavicle
* pathological fracture
* patient is unable to medically tolerate general anesthesia
* patient is unable to provide informed consent or comply with completing questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated surgically for diaphysial clavicle fracture.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Functional outcome as measured by Constant Shoulder Score and Disabilities of the Arm, Shoulder and Hand (DASH) score | 1+ year post-op
  The primary outcome measure for this study will be incision related numbness, based on clinical examination and the use of our skin numbness map. Our null hypothesis is that there will be no difference in incision related numbness between the two groups: percutaneous versus open approach. Our primary objective is to disprove this hypothesis, predicting that the percutaneously treated group will have less incisional numbness.

SECONDARY OUTCOMES:
Incision numbness at surgical site. | 2 wks, 6 wks, 3 mths, 6mnths and 1+ year post-op
  Our secondary outcome measures will be union, malunion, and nonunion rates between these two methods, as well as infection rates and functional and satisfaction outcomes based on subjective questioning and the DASH and Constant shoulder score questionnaires. Our null hypothesis for these secondary outcomes is that there will be no difference between the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Kubiak, MD, Principal Investigator — University of Utah; Thomas Christensen, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopedic Center, Salt Lake City, Utah, United States